CLINICAL TRIAL: NCT05632380
Title: The Safety and Efficacy of Autologous Hematopoietic Stem Cell Transplantation (ASCT) in Combination With C-CAR088, an Autologous BCMA CAR-T Cell Product, for Treating Patients With Ultra High-risk Multiple Myeloma
Brief Title: ASCT in Combination With C-CAR088 for Treating Patients With Ultra High-risk Multiple Myeloma (MM)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022012
Record Dates: First submitted 2022-11-08; First posted 2022-11-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASCT and C-CAR088 (Experimental): Patients will undergo ASCT followed by C-CAR088 single dose infusion.
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation; Biological: C-CAR088

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation — Patients receive transplantation conditioning followed by autologous hematopoietic stem cell transplantation after successful stem cell mobilization and collection. If previously collected stem cells are available, no stem cell mobilization or collection is required, and patients will receive conditioning directly.
Biological: C-CAR088 — C-CAR088 is an BCMA targeted Chimeric Antigen Receptor-T cell product. Patients will receive C-CAR088 single dose infusion 3 days after ASCT. The dose level of C-CAR088 will be determined by the investigator.

SUMMARY:
This is a phase I/II, single-arm, open-lable study of autologous stem cell transplantation in combination with C-CAR088, an autologous BCMA CAR-T cell product, for patients with ulta high-risk multiple myeloma, defined as failed or unsatisfied responses to front line VRD-based treatment with or without the presence of multiple high-risk cytogenetic features.

DETAILED DESCRIPTION:
Patients with ultra high-risk multiple myeloma will undergo leukapheresis, stem cell mobilization and collection (could omit if collected before screening), conditioning, ASCT and C-CAR088 infusion. Patients receive a single dose of C-CAR088 three days post-ASCT. Two conditioning protocols and two dose levels of C-CAR088 will be used based on the investigator's discretion. Patients will be evaluated closely for safety of efficacy during the first three months, then less frequently in the following months until 24 months post-ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Transplantation eligible patients, male or female, aged 18 to 65 years
* Ultra high risk multiple myeloma, defined as failed or unsatisfied responses to front line VRD-based treatment with or without the presence of multiple high-risk cytogenetic features
* Adequate liver, renal, bone marrow, and heart function
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-1.
* Male and female of reproductive potential must agree to use birth control during the study.

Exclusion Criteria:

* Known allergies to the components or excipients of the C-CAR088 cell product
* Prior allogenic HSCT, or ASCT
* CNS involvement
* Stroke or convulsion history within 6 months prior to signing ICF
* Autoimmune disease, immunodeficiency or disease requiring immunosuppressants treatment
* Uncontrolled active infection; active HBV, HCV infection; HIV or syphilis Infection
* Severe heart, liver, renal or metabolism disease
* Inadequate wash-out time for previous anti-tumor treatments prior to apheresis
* Previous CAR-T cell treatment, genetically modified T-cell therapies or BCMA-directed treatment history
* History or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's safe participation and compliance in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and severity of adverse events (AE) | 24 months
  Incidence rate and severity of adverse events (AE)

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 months
  The time from the initiation of study treatment to the date of first documented disease progression or death
MRD negativity rate | 24 months
  The percentage of patients who reached MRD negativity
Overall response rate (ORR) | 24 months
  The percentage of patients who reached PR, VGPR, CR or sCR as their best response
Duration of response (DOR) | 24 months
  The time from the first documented PR or better response to progression or death, whichever occurs first
Time to response (TTR) | 24 months
  The time between the initiation of study treatment until the the first documented PR or better response
Overall Survival (OS) | 24 months
  OS is defined as the time from the initiation of study treatment to death from any cause
Cmax (maximal plasma concentration) | 24 months
  Maximal plasma concentration of C-CAR088 in peripheral blood
Tmax (Time to reach the maximal plasma conceration) | 24 months
  Time to reach the maximal plasma conceration of C-CAR088 in peripheral blood
AUC0-28d (area under the curve from day 0-day 28) | 28 days post C-CAR088 infusion
  Area under the curve of C-CAR088 in peripheral blood within 28 days post C-CAR088 infusion
Tlast (Time of last measurable observed concentration) | 24 months
  Time of last measurable observed concentration of C-CAR088 in peripheral blood

OTHER OUTCOMES:
Anti-drug (C-CAR088) antibody | 24 months
  The correlation between the presence of anti-drug (C-CAR088) antibody with the efficacy and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, M.D., PH.D., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China